CLINICAL TRIAL: NCT02389517
Title: Phase II Randomized Trial of Continuation of Post-Transplant Maintenance With Single-Agent Lenalidomide vs. Consolidation/Maintenance With Ixazomib-Lenalidomide-Dexamethasone in Patients With Residual Myeloma
Brief Title: Lenalidomide With or Without Ixazomib Citrate and Dexamethasone in Treating Patients With Residual Multiple Myeloma After Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Multiple Myeloma Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-0899; NCI-2015-00138 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); X16047; 14-0899; IRB14-0899 (Other: University of Chicago); P30CA014599 (NIH)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Plasma Cell Myeloma; Residual Disease
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual | interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (ixazomib citrate, lenalidomide, dexamethasone) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, and 15, lenalidomide PO QD on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22 (of courses 1-4 only).
  Interventions: Drug: Ixazomib Citrate; Drug: Lenalidomide; Drug: Dexamethasone
- Arm II (lenalidomide) (Active Comparator): Patients receive lenalidomide PO as in Arm I.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; proteasome inhibitor MLN9708
  Arms: Arm I (ixazomib citrate, lenalidomide, dexamethasone)
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; IMiD-1
Drug: Dexamethasone — Given PO
  Other Names: DM
  Arms: Arm I (ixazomib citrate, lenalidomide, dexamethasone)

SUMMARY:
This randomized phase II trial studies how well lenalidomide alone compared to lenalidomide, ixazomib citrate, and dexamethasone work in treating patients with multiple myeloma that remains (residual) after donor stem cell transplant. Lenalidomide may help the immune system kill abnormal blood cells or cancer cells and may also prevent the growth of new blood vessels that are needed for cancer growth. Ixazomib citrate may stop the growth of cancer cells by interfering with proteins necessary for cell growth. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether lenalidomide is more effective with or without ixazomib citrate and dexamethasone in treating residual multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of minimal residual disease (MRD)-negative disease by multiparameter-flow cytometry at 12 months after randomization.

SECONDARY OBJECTIVES:

I. Evidence of response as demonstrated by the improvement of the depth of response by at least one category according to International Myeloma Working Group (IMWG) response criteria.

II. Progression free survival (PFS). III. Overall survival (OS). IV. Duration of MRD-negative disease. V. Safety and tolerability of experimental arm (ixazomib citrate, lenalidomide, and low dose dexamethasone [IRd]) vs. control arm (lenalidomide [Rd]).

TERTIARY OBJECTIVES:

I. Determination of markers of response based on pre-treatment characteristics using methods described in correlative research.

II. Evaluation of MRD by gene sequencing method using the Sequenta platform (LymphoSIGHT®) in parallel with multi-parameter flow cytometry (MFC).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive ixazomib citrate orally (PO) on days 1, 8, and 15, lenalidomide PO once daily (QD) on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22 (of courses 1-4 only).

ARM II: Patients receive lenalidomide PO as in Arm I.

In both arms, treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After the completion of treatment, patients are followed up at 30 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed induction treatment followed by autologous stem cell transplant as initial therapy for symptomatic myeloma as per IMWG criteria and initiated Revlimid (lenalidomide) maintenance

  * Patients must have initiated lenalidomide maintenance at approximately 3 months post autologous stem transplant (preferably 70-90 but not more than 120 days)
  * Patients must be receiving lenalidomide 10 mg or 15 mg and be able to tolerate dose escalation to 25 mg daily
  * Patients must have received lenalidomide maintenance for 3 months (+1 month window for a maximum of 4 months lenalidomide prior to enrollment)
* No evidence of progressive disease on lenalidomide
* Any measurable residual disease at the time of screening for the study documented in at least one of the following ways:

  * Serum protein electrophoresis (SPEP)/immunofixation studies (IFIX) positive disease
  * Freelite only positive disease
  * SPEP/IFIX - negative and Freelite- negative but MRD-positive disease is allowed
* Evidence of MRD at the time of screening for this study by multi-color flow cytometry (bone marrow procedure at screening required)
* Bone marrow specimen will be required at study entry; available deoxyribonucleic acid (DNA) sample will be used for calibration step for MRD evaluation by gene sequencing
* Life expectancy of more than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Bilirubin =<1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Hemoglobin >= 8 g/dL
* Platelet count >= 75 x 10^9/L
* Calculated creatinine clearance (by Cockroft-Gault) >= 50 ml/min or serum creatinine below 2 g/dL
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)

Exclusion Criteria:

* Evidence of progressive disease on lenalidomide maintenance as per IMWG criteria
* Patients who have already started or received multi-drug consolidation regimen post-transplant expect for lenalidomide maintenance
* Diarrhea > grade 1 in the absence of anti-diarrheals
* Central nervous system involvement
* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* History of allergy to mannitol
* Major surgery within 14 days before enrollment
* Radiotherapy within 14 days before randomization; if the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled cardiac conditions such as hypertension, or cardiac arrhythmias, or New York Heart Association stage III and IV congestive heart failure, or unstable angina or myocardial infarction within the past 6 months
* Rate-corrected QT interval of electrocardiograph (QTc) > 470 msec on a 12-lead electrocardiogram (ECG) during screening
* Uncontrolled diabetes
* Acute infection requiring systemic anti-infectives, antivirals, or antifungals within two weeks prior to first dose
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong inhibitors of cytochrome P450 family 3, subfamily A, polypeptide 2 (CYP1A2) (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P450 family 3, subfamily A CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease; patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patient has >= grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2024-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Jakubowiak, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) | Arm II (Lenalidomide)
Started | 20 | 22
Completed | 14 | 17
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Progressive disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) | Arm II (Lenalidomide) | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Full Range); unit: years] | 62.6 [43.7 to 73.4] | 59.1 [38.6 to 74.3] | 60.8 [38.6 to 74.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 14 | 16 | 30
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With MRD Negativity
Description: Rate of MRD negativity after 12 months of treatment with Ixazomib in combination with lenalidomide and dexamethasone compared to MRD negativity rate after 12 months of lenalidomide alone. For the majority of patients, where MRD positivity at screening will be determined by Multi-parameter Flow Cytometry (MFC), an improvement will be defined as a conversion from MRD-positive to MRD-negative disease by MFC. Additionally, in the fraction of patients with MRD-negative disease by MFC at screening, who were MRD-positive by Next Generation Sequencing (NGS), an improvement will be defined as a conversion from MRD-positive to MRD-negative disease by NGS
Time Frame: At 12 months
Population: The data for 3 patients in Arm 1 AND 4 patients in Arm II were not collected.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) | Arm II (Lenalidomide)
Number analyzed (Participants) | 11 | 13
percentage of participants | 18 | 31

2. Secondary Outcome: Overall Response (Number of Participants With VGPR, CR, sCR)
Description: Overall response was defined according to IMWG criteria as
  1. very good partial response (VGPR)
  2. complete response (CR)
  3. stringent complete response (sCR)
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) | Arm II (Lenalidomide)
Number analyzed (Participants) | 14 | 17
Participants
  VGPR | 5 | 3
  CR | 5 | 6
  sCR | 2 | 0

3. Secondary Outcome: Duration of MRD-negative Disease
Description: Duraion of MRD-negativie disease was defined as the duration from the date of MRD negative to the date of diseae progression or date of last clinical follow up.
Time Frame: every 28 days, up to 2 years
Population: Patients who had MRD-negative were analyzed.
Measure: Median (Full Range); unit: years
Arm/Group | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) | Arm II (Lenalidomide)
Number analyzed (Participants) | 2 | 4
years | 1.91 [1.84 to 1.98] | 1.98 [1.82 to 2.0]

4. Secondary Outcome: Progression Free Survival
Description: Time to event will be estimated using the product-limit method of Kaplan and Meier.
Time Frame: up to 2 years
Population: One patient in Arm1 and two patients in Arm 2 were not analyzed because their data were not collected.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) | Arm II (Lenalidomide)
Number analyzed (Participants) | 19 | 20
years | NA [2.2 to NA] — Insufficient number of participants with events to calculate via KM methodology | NA [NA to NA] — Insufficient number of participants with events to calculate via KM methodology

5. Secondary Outcome: Overall Survival
Description: OS is the time from randomization date to death date. Participants who have not died will be censored on the last date they are known to be alive.
Time Frame: Up to 2 years
Population: One patients in Arm 1 and two patients in Arm 2 were not analyzed because their data were not collected.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) | Arm II (Lenalidomide)
Number analyzed (Participants) | 19 | 20
years | NA [NA to NA] — Median and 95% Confidence Interval could not be calculated due to an insufficient number of participants with events | NA [NA to NA] — Median and 95% Confidence Interval could not be calculated due to an insufficient number of participants with events

6. Secondary Outcome: Number of Patients With Adverse Events
Description: Graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Up to 30 days post-treatment, **up to 2 years**
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) | Arm II (Lenalidomide)
Number analyzed (Participants) | 20 | 22
Participants
  Abdominal pain | 2 | 1
  Agitation | 2 | 0
  Alanine aminotransferase increased | 1 | 2
  Allergic reaction | 1 | 0
  Allergic rhinitis | 1 | 1
  Anemia | 1 | 4
  Anorexia | 1 | 0
  Anxiety | 2 | 0
  Arthraigia | 1 | 3
  Aspartate aminotransferase increased | 1 | 1
  Back Pain | 5 | 5
  Bloating | 3 | 2
  Blurred vision | 2 | 1
  Bronchospasm | 1 | 0
  Bruising | 5 | 1
  Buttock pain | 1 | 0
  Chills | 1 | 0
  Confusion | 2 | 1
  Conspipation | 7 | 5
  Cough | 6 | 4
  Dehydration | 1 | 0
  Depression | 4 | 1
  Diarrhea | 19 | 11
  Dizziness | 3 | 5
  Dry eye | 1 | 1
  Dry mouth | 2 | 0
  Dysgeusia | 1 | 1
  Dyspepsia | 1 | 1
  Dyspnea | 4 | 4
  Ear pain | 1 | 1
  Edema Limbs | 6 | 3
  Edema trunk | 1 | 0
  Eye disorders - others | 2 | 1
  Fall | 1 | 1
  Fatigue | 10 | 9
  Fever | 3 | 3
  Flu like symptoms | 4 | 5
  Flushing | 2 | 0
  Fracture | 1 | 0
  Gait disturbance | 1 | 0
  Generalized muscle weakness | 2 | 0
  Gum infection | 1 | 0
  Headache | 3 | 1
  Hypertension | 1 | 0
  Hypokalemia | 3 | 3
  Hypomagnesemia | 1 | 1
  Hyponatremia | 1 | 0
  Hypotension | 1 | 0
  Hypoxia | 1 | 0
  Immune system disorders | 1 | 0
  Infections and infestations | 3 | 2
  INR increased | 1 | 0
  Insomnia | 6 | 0
  Irritability | 2 | 0
  Joint range of motion decreased cervical spine | 1 | 0
  Lethargy | 1 | 0
  Leukocytosis | 1 | 0
  Libido decreased | 1 | 0
  Localized edema | 1 | 1
  Lung infection | 1 | 3
  Lymphocyte count decreased | 2 | 0
  Memory impariment | 1 | 0
  Metabolism and nutrition disorders - Other, specify | 1 | 0
  Mucosal infection | 1 | 0
  Mucositis oral | 3 | 0
  Muscle weakness lower limb | 1 | 0
  Muscle weakness upper limb | 2 | 0
  Myalgia | 4 | 4
  Nasal congestion | 2 | 3
  Nausea | 10 | 4
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify | 1 | 1
  Neutrophil count decreased | 7 | 5
  non-cardiac chest pain | 1 | 0
  Oral dysesthesia | 1 | 0
  Oral pain | 1 | 0
  Otitis externa | 1 | 0
  Pain | 4 | 5
  Pain in extremity | 5 | 2
  Papulopustular rash | 2 | 1
  Paresthesia | 1 | 1
  Paronychia | 1 | 0
  Peripheral motor neuropathy | 1 | 1
  Peripheral sensory neuropathy | 5 | 5
  Platelet count decreased | 7 | 2
  Psychiatric disorders - Other, specify | 1 | 0
  Rash maculo-papular | 3 | 1
  Renal and urinary disorders - Other, specify | 1 | 0
  Sepsis | 2 | 0
  Sinus bradycardia | 1 | 1
  Skin and subcutaneous tissue disorders - Other, specify | 4 | 2
  skin hyperpigmentation | 1 | 0
  Small intestine infection | 1 | 0
  Sore throat | 3 | 1
  Spasticity | 2 | 0
  Syncope | 1 | 1
  Tinnitus | 2 | 1
  Tooth infection | 1 | 0
  Toothache | 1 | 0
  Tremor | 4 | 0
  Upper respiratory infection | 7 | 6
  Urinary frequency | 3 | 0
  Urinary incontinence | 1 | 0
  Urinary retention | 1 | 0
  Urinary tract infection | 2 | 0
  Vaginal discharge | 1 | 0
  Vascular disorders - Other, specify | 1 | 0
  Vomiting | 6 | 1
  Weight gain | 2 | 1
  Wheezing | 1 | 0
  White blood cell decreased | 1 | 1
  Acute kidney injury | 0 | 1
  Anal pain | 0 | 1
  Bone pain | 0 | 1
  Bronchial Infection | 0 | 1
  Cardiac disorders - Other, specify | 0 | 1
  chest pain -cardiac | 0 | 1
  Conjunctivitis | 0 | 1
  Creatinine Increased | 0 | 2
  Cystitis noninfective | 0 | 1
  Dry skin | 0 | 2
  External ear inflammation | 0 | 1
  Flank pain | 0 | 1
  Gastroesophageal reflux disease | 0 | 1
  Gastrointestinal disorders - Other, specify | 0 | 1
  Gingival pain | 0 | 1
  Hyperglycemia | 0 | 1
  Hearing impaired | 0 | 2
  Hemorrhoidal hemorrhage | 0 | 1
  Hypocalcemia | 0 | 3
  Hypophosphatemia | 0 | 1
  Musculoskeletal and connective tissue disorder - Other, specify | 1 | 3
  Neck pain | 0 | 3
  Personality change | 0 | 1
  Postnasal drip | 0 | 2
  Pruritus | 0 | 2
  Rash aceniform | 0 | 1
  Respiratory, thoracic and mediastinal disorders - Other, specify | 0 | 4
  Sinus tachycardia | 0 | 1
  Sinusitis | 0 | 1
  Somnolence | 0 | 1
  Superficial thrombophlebitis | 0 | 1
  Supraventricular tachycardia | 0 | 1
  Thromboembolic event | 0 | 1
  Vertigo | 0 | 2
  Weight loss | 0 | 1

7. Secondary Outcome: Overall Response (Number of Participants With VGPR, CR, sCR)
Description: as for outcome 2
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) | Arm II (Lenalidomide)
Number analyzed (Participants) | 14 | 17
Participants
  VGPR | 3 | 6
  CR | 5 | 5
  sCR | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years after the end of treatment visit, ** up to 2.5 years**
Arm/Group | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) | Arm II (Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 5/20 | 2/22
Other Adverse Events (participants affected / at risk) | 20/20 | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) (N=20) | Arm II (Lenalidomide) (N=22)
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fever (General disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infections and infestations - others (Infections and infestations) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Neoplasms benign, malignant and unspecified - others (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory, thoracic and mediastinal disorders- others (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Ixazomib Citrate, Lenalidomide, Dexamethasone) (N=20) | Arm II (Lenalidomide) (N=22)
abdominal pain (Gastrointestinal disorders) | 2 | 1
Agitation (Psychiatric disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2
Allergic reaction (Immune system disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 4
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Bloating (Gastrointestinal disorders) | 3 | 2
Blurred vision (Eye disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 5 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardiac disorders - others (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 1
Conjuinctivitis (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Creatinine increased (Investigations) | 0 | 2
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 4 | 1
Diarrhea (Gastrointestinal disorders) | 19 | 11
Dizziness (Nervous system disorders) | 3 | 5
Dry eye (Eye disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Ear pain (Ear and labyrinth disorders) | 1 | 1
Edema limbs (General disorders) | 6 | 3
Edema trunk (General disorders) | 1 | 0
Eye disorders- others (Eye disorders) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fatigue (General disorders) | 10 | 9
Fever (General disorders) | 3 | 3
Flu like symptoms (General disorders) | 4 | 5
Flushing (Vascular disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Gum infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Immune system disorders- others (Immune system disorders) | 1 | 0
Infections and infestations-other (Infections and infestations) | 2 | 2
INR increased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 6 | 0
Irritability (General disorders) | 2 | 0
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 1
Localized edema (General disorders) | 1 | 1
Lung infection (Infections and infestations) | 1 | 2
Lymphocyte count decreased (Investigations) | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Metabolism and nutrition disorders - other (Metabolism and nutrition disorders) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal and connective tissue disorder-other (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 10 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Neoplasms benign, malignant and unspecified - other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutrophil count decreased (Investigations) | 7 | 5
Non-cardiac chest pain (General disorders) | 1 | 0
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Pain (General disorders) | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Populopustular rash (Infections and infestations) | 2 | 1
Paresthesia (Nervous system disorders) | 1 | 1
Paronychia (Infections and infestations) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 5
Platelet count decreased (Investigations) | 7 | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruitus (Skin and subcutaneous tissue disorders) | 0 | 2
Psychiatric disorders-other (Psychiatric disorders) | 1 | 0
Renal and urinary disorders-other (Renal and urinary disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders-other (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Sinus bradycardia (Cardiac disorders) | 1 | 1
Skin and subcutaneous tissue disorders-other (Skin and subcutaneous tissue disorders) | 4 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Small intestine infection (Infections and infestations) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Spasticity (Nervous system disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Tooth infection (Infections and infestations) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Tremor (Nervous system disorders) | 4 | 0
Upper respiratory infection (Infections and infestations) | 6 | 6
Urinary frequency (Renal and urinary disorders) | 3 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vascular disorders-other (Vascular disorders) | 1 | 0
Vertigo (Gastrointestinal disorders) | 0 | 2
Weight gain (Investigations) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT02389517/Prot_SAP_000.pdf